CLINICAL TRIAL: NCT05080569
Title: LUMO Study: Luteal Phase Support in IUI MOH Treatment Luteal Phase Support in IUI MOH
Brief Title: Luteal Phase Support in IUI MOH Treatment Luteal Phase Support in IUI MOH Treatment
Acronym: LUMO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Frank JM Broekmans, Professor in Reproductive Endocrinology & Surgery, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2359660
Record Dates: First submitted 2021-08-09; First posted 2021-10-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy Related; Fertility Issues; Luteal Phase Defect; Infertility Unexplained
Keywords: progesterone; Cost-effective; Intrauterine insemination; live birth; luteal support; ongoing pregnancy; ovulation induction; unexplained infertility
MeSH Terms: conditions — Infertility | interventions — Utrogestan

STUDY DESIGN:
Intervention Model Description: The LUMO study is a multicenter, randomized, placebo-controlled trial with cost-effectiveness analysis. Participating sites consist of academic and non-academic hospitals and fertility clinics. There are two treatment arms (MOH/IUI treatment with LPS vs MOH/IUI treatment with placebo) with a non-blinded superiority design. Participants are randomly distributed across both treatment arms for the entire study-period (six months, non-crossover).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded superiority design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOH/IUI treatment with LPS (Experimental): (Mild) Ovarian stimulating treatment and insemination are according to regular treatment protocol. Females assigned to the treatment group start LPS, applying 3dd200mg Utrogestan in vaginal capsules, on the day of IUI. Treatment is continued until the onset of menstruation, a negative pregnancy test, miscarriage or confirmed vital intra-uterine pregnancy at 7 weeks gestation
  Interventions: Drug: Progesterone Vaginal Product
- MOH/IUI treatment with placebo (Placebo Comparator): Females will receive regular MOH/IUI treatment. The female cycle is mildly stimulated and monitored until the desired amount of ripe follicles is achieved. In the absence of other reasons to cancel the treatment, ovulation is triggered and subsequently pre-washed semen is inseminated into the uterus.
  Females assigned to the placebo group start placebo, applying 3dd1 vaginal capsules, on the day of IUI. Treatment is continued until the onset of menstruation, a negative pregnancy test, miscarriage or confirmed vital intra-uterine pregnancy at 7 weeks gestation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone Vaginal Product — 3dd200mg
  Other Names: Utrogestan
  Arms: MOH/IUI treatment with LPS
Drug: Placebo — 3dd1 vaginal capsule
  Arms: MOH/IUI treatment with placebo

SUMMARY:
The LUMO study is a multicenter, randomized controlled trial that evaluates the effectivity of luteal phase support in MOH/IUI treatment.

DETAILED DESCRIPTION:
Participating sites consist of academic and non-academic hospitals and fertility clinics in The Netherlands. There are two treatment arms (MOH/IUI treatment with LPS vs MOH/IUI treatment with placebo) with a non-blinded superiority design. Participants are randomly distributed across both treatment arms for the entire study-period (six months, non-crossover).

Eligibility criteria are: 1) couples starting IUI with Mild Ovarian HyperStimulation (MOH), with the intend to receive this treatment for at least six months. 2) Indication for MOH/IUI treatment is in accordance with current (dutch) NVOG guidelines; Diagnosis of unexplained (primary or secondary) infertility with Hunault <30% (or >30%, after an expectant management period of at least 6 additional months). Total mobile sperm count (VCM) >10 million. 3) Females aged >18 years with regular menstrual cycle.

(Mild) Ovarian stimulating treatment and insemination are according to regular treatment protocol. Females assigned to the treatment group start LPS, applying 3dd200mg Utrogestan in vaginal capsules, on the day of IUI. Treatment is continued until the onset of menstruation, a negative pregnancy test, miscarriage or confirmed vital intra-uterine pregnancy at 7 weeks gestation.

Main outcome is pregnancy within 6 months of treatment, leading to Live birth. Secondary outcomes are; Clinical pregnancy rate. Miscarriage rate. Multiple pregnancy rate. Pregnancy complications. Perinatal outcomes. Side effects and compliance to therapy. Added Medication Costs. Budget impact.

The analyses will include a cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Couples starting IUI with Mild Ovarian HyperStimulation (MOH), with the intend to receive this treatment for at least six months.
* Diagnosis of unexplained (primary or secondary) infertility
* Hunault <30% (or >30%, after an expectant management period of at least 6 additional months).
* Females aged >18 years with regular menstrual cycle.
* Total mobile sperm count (VCM) >10 million.

Exclusion cirteria:

* Cycle irregularities
* Male factor infertility

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1008 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Live Birth | 6 months
  Pregnancy leading to Live birth within six months.

SECONDARY OUTCOMES:
Clinical pregnancy rate | <6 months
  Number and rate of patients that achieve a clinical pregnancy within six months
Miscarriage rate | <6 months
  Number and rate of patients that experience miscarriage (gestation <16weeks) within six months
Multiple pregnancy rate | <6 months
  Number of pregnancies with 2 or more fetuses
Pregnancy complications | 1 year
  Pregnancies complicated by preterm labor (<37 weeks), loss of pregnancy (>16weeks), gestational diabetes, preeclampsia, HELLP syndrome or pregnancy induced hypertension.
Perinatal outcomes | <6 weeks
  Stillbirth/Livebirth/Perinatal death, Gestational age at delivery, birthweight
Side effects | <1 year
  Nausea, stomach ache, vaginal discharge, other (self reported) side effects
Compliance to therapy | 6 months
  Use of medication as prescribed
Added medication costs | 1 year
  Increae in total therapy costs due to the addition of Utrogestan (the treatment).
Budget impact | 1 year
  Economic assessment that estimated financial consequences of adopting a new intervention

CONTACTS AND LOCATIONS:
Overall Officials: Broekmans, Prof. Dr., Principal Investigator — Professor Reproductive Medicine
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
After finishing the project, data will not be shared publicly, but under restricted access, as the data is privacy sensitive. We publish the descriptive metadata in the data repository with a description of how a data request can be made (by sending an email to the corresponding author). If other researchers like to reuse our data, this can only be granted if the research question is in line with the original informed consent signed by the study participants. Every application therefore will be screened upon this requirement. If granted, a data usage and transfer agreement is signed by the receiving party. The specific data that will be shared with third parties after approval of the Principal Investigator, will be determined on a case-by case basis. Based on the specific research question, all raw data including the codebook and scripts of analysis in SPSS/R may be shared if considered of added value and with mutual trust and agreement in a Data usage agreement.

REFERENCES:
- [Derived] Preesman E, Drechsel K, Crommelin H, Broekmans F, Verpoest W, Broer S; LUMO Study Group. Does luteal phase support in MOH-IUI treatment improve cumulative live birth rates in couples with unexplained subfertility? Study protocol of the LUMO study: a centre, randomised, double-blind, controlled trial with cost-effectiveness analysis. BMJ Open. 2025 Nov 19;15(11):e111872. doi: 10.1136/bmjopen-2025-111872. PMID 41263858